CLINICAL TRIAL: NCT00184132
Title: The Effects of Different Interior Decorations in a Psychiatric Intensive Care Unit.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); County of South Trøndelag (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEV-00
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Mental Disorders
Keywords: Intensive care units; Emergency services, psychiatric; Interior Design and Furnishings; Intensive Care
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norwegian home style ward (Experimental): The walls received wainscots, colourful wallpaper and paintings; the ceilings were lowered and had multiple lighting spots, the windows tasteful curtains; we put wardrobes, chairs, flowers and personal items in the patient rooms; and Italian ceramic tile covered the entire bathroom
  Interventions: Procedure: Psychiatric intensive care unit in Norwegian home style
- sparsely furnished ward (Active Comparator): traditional interior design and furnishings. The rooms had sparse furniture, walls in grey colours lacking pictures, no window curtains, single lamps in the ceiling 4 m high, bathroom with grey, laminated paint all over, and patient rooms with a single bed and a chair of metal tubes
  Interventions: Procedure: Psychiatric intensive care unit sparsely furnished and not decorated

INTERVENTIONS:
Procedure: Psychiatric intensive care unit in Norwegian home style
  Arms: Norwegian home style ward
Procedure: Psychiatric intensive care unit sparsely furnished and not decorated
  Arms: sparsely furnished ward

SUMMARY:
The purpose of the study is to compare effects of treatment of patients acutely admitted to a Psychiatric Intensive Care Unit (PICU) with either a sparsely decorated interior or interior decorations like an ordinary, Norwegian home.

DETAILED DESCRIPTION:
The PICU in Østmarka psychiatric department, St. Olavs Hospital contains 2 identical parts. Each part contains 2 beds. The PICU had a traditional sparsely decorated interior. In cooperation with architects and the county building authorities one of the parts were redecorated to an interior like an ordinary Norwegian home. All patients admitted the the PICU were semi-randomized to either traditional or "Norwegian home" interior decorations. Symptoms, behaviour, and treatment were evaluated at admittance, day 3 and discharge from the PICU

ELIGIBILITY:
Inclusion Criteria:

* All patients acutely admitted to the PICU, St. Olavs Hospital, Østmarka dep.

Exclusion Criteria:

* Patients with dementia or mental retardation to an extensive degree.
* Patients not speaking Norwegian or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2000-11 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Length of stay in days | 1 month
Scores on general psychiatric rating scale | 3 days
  Positive and Negative Syndrome Scale (PANSS)
Scores on violent or threatening incidents | 3 days
  recorded with Staff Observation Aggression ScaleRevised (SOAS-R)

SECONDARY OUTCOMES:
Therapeutic steps daily | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Olav M Linaker, Professor, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Østmarka Psychiatric Department, St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vaaler AE, Morken G, Linaker OM. Effects of different interior decorations in the seclusion area of a psychiatric acute ward. Nord J Psychiatry. 2005;59(1):19-24. doi: 10.1080/08039480510018887. PMID 16195094
- [Derived] Vaaler AE, Iversen VC, Morken G, Flovig JC, Palmstierna T, Linaker OM. Short-term prediction of threatening and violent behaviour in an Acute Psychiatric Intensive Care Unit based on patient and environment characteristics. BMC Psychiatry. 2011 Mar 18;11:44. doi: 10.1186/1471-244X-11-44. PMID 21418581
- [Derived] Flovig JC, Vaaler AE, Morken G. Effects of legal and illegal use of benzodiazepines at acute admission to a psychiatric acute department. BMC Res Notes. 2010 Oct 19;3:263. doi: 10.1186/1756-0500-3-263. PMID 20958975